CLINICAL TRIAL: NCT01247623
Title: Trial With Telomerase Peptide Vaccine In Combination With Temozolomide in Patients With Advanced Malignant Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Other Study IDs: P03700
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Malignant Melanoma
Keywords: Non-resectable, advanced malignant melanoma.
MeSH Terms: conditions — Melanoma | interventions — GV1001 peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: GV1001

SUMMARY:
Primary objective: Determination of safety and tolerability of GV1001 administration combined with Temozolomide (based on blood samples and adverse events).

Feasibility of combining active immunisation with Temozolomide treatment. Determination of immunological response after administration of GV1001 and Temozolomide as measured by presence of DTH skin test reaction and specific T-cell responses.

Secondary: Evaluation of objective tumour response

The trial is an exploratory study which main objective is to estimate safety and feasibility of combining active immunisation with chemotherapy. However, the trial may also indicate the efficacy of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of malignant melanoma.
* Previously untreated and non-resectable disease
* Measurable or evaluable tumour.
* Age ≥ 18 and ≤ 75 years.
* Performance status ECOG-WHO 0, 1 and 2 (Appendix III)
* Written informed consent (Appendix II)
* Adequate bone marrow liver, heart and renal function:
* WBC count >3.0 x 109/L and platelets count >100 x 109/L.
* ASAT, ALAT <2 x upper normal laboratory value.
* Serum creatinine <2 x upper normal laboratory value.

Exclusion Criteria:

* Previous treatment with chemotherapy.
* Clinical signs of brain metastases.
* Severe cardiac insufficiency (NYHA III or IV) with uncontrolled and/or unstable cardiac or coronary artery disease.
* Severe active infections such as HIV or hepatitis B or Hepatitis C.
* Medication for severe intercurrent disease which might affect immunocompetence (e.g. immunosuppressants, systemic corticosteroids).
* Pregnancy, breast-feeding or absence of adequate contraception for fertile patients.
* Simultaneously participation in other clinical studies.
* Any reason why, in the opinion of the investigator, the patient should not participate.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Postbox 4953, Norway